CLINICAL TRIAL: NCT01346462
Title: A Randomized Controlled Trial of a Novel Community Health Worker Care Transitions Intervention.
Brief Title: IMPaCT (Individualized Management Towards Patient-Centered Targets)
Acronym: PaCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Shreya Kangovi, Philadelphia Veterans Affairs Medical Center Special Fellow, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB 813426
Record Dates: First submitted 2011-04-29; First posted 2011-05-03 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: General Medical Inpatient Conditions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PaCT (Experimental): The Patient-Centered Transition Arm
  Interventions: Behavioral: Patient-Centered Transition Intervention
- Control (No Intervention): Control group patients will receive routine care from the admitting hospital, including routine patient management, and discharge planning.

INTERVENTIONS:
Behavioral: Patient-Centered Transition Intervention — Community Health Workers will act as PaCT Partners for uninsured/Medicaid patients who are being discharged from the Hospital of the University of Pennsylvania and Presbyterian Hospital. PaCT Partners will help patients to overcome the challenges of transition, including arranging primary care provider (PCP) follow-up, filling medication prescriptions and obtaining referrals to community-based social services.
  Arms: PaCT

SUMMARY:
The investigators propose a pilot randomized controlled trial of a care transitions intervention in which trained Community Health Workers will act as supports for socioeconomically vulnerable patients who are being discharged from the Hospital of the University of Pennsylvania and Presbyterian Hospital. CHWs or IMPaCT Partners will help patients to overcome the challenges of transition, including arranging primary care provider (PCP) follow-up, filling medication prescriptions and obtaining referrals to community-based social services. As our primary outcome, the investigators will examine the effect of the IMPaCT intervention on rates of primary care follow-up. The investigators will also examine the effect of IMPaCT on secondary outcome variables including patients' satisfaction with the experience of transition, quality of discharge communication, medication adherence, self- rated health, and inpatient readmission within 30 days after discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Participant admitted to the General Medicine services of the Hospital of the University of Pennsylvania (HUP), or Presbyterian Hospital during the enrollment period
2. Participant uninsured or insured by Medicaid at the time of discharge from the hospital
3. Participant is 18-65 years old
4. Participant is willing to participate and be contacted at 14 days post-discharge by telephone or through a home visit by research personnel (if no functioning telephone is present in the household)
5. Participant resides in one of the following zip codes: 19104, 19131, 19139, 19143, 19146. These zip codes have the highest frequency of readmissions to HUP and Presbyterian Hospital
6. Participant is English speaking

Exclusion Criteria:

1. Patients with insurance other than Medicaid will be excluded as they are outside of the population of interest for this intervention targeted specifically at socioeconomically vulnerable patients. Dual eligible patients (Medicaid and Medicare) will be excluded. Patients older than 65 are eligible for the Transitional Care Model Intervention, which is a separate intervention offered at Penn Medicine hospitals.
2. Non-English speaking participants will be excluded because in this pilot study, the study only has English-speaking PaCT personnel. In future studies, it will be important to study the effect of PaCT in non-English speaking populations.
3. Patients outside of the target zipcodes are being excluded for feasibility reasons during this pilot study: with only two PaCT Partners, we are choosing to focus our resources on a geographic area that has the highest rates of readmissions in order to facilitate home visits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Completion of Follow-up Appointment with PCP | 14 days post discharge
  We hypothesize that compared to patients who receive usual discharge planning, PaCT patients will have a higher proportion of follow-up to PCP within two weeks post-discharge, compared with usual discharge planning.

SECONDARY OUTCOMES:
Morisky Medication Adherence scale. | 14 days post-discharge
  We hypothesize that compared to patients with usual discharge planning, PaCT patients will have higher medication adherence as measured by the Morisky Medication Adherence scale.
Patient Activation Measure | 14 days post discharge
  We hypothesize that compared to patients with usual discharge planning, PaCT patients will exhibit a higher level of patient activation as measured by the Patient Activation Measure.
Self-rated Health | 14 days post-discharge
  We hypothesize that compared with usual discharge planning, PaCT patients will report better health as measured by the Short Form Health Survey (SF-12) at 14 days post-discharge.
Patient Satisfaction Questionnaire | 14 days post discharge
  We hypothesize that compared with usual discharge planning, PaCT patients will report higher satisfaction as measured by the Patient Satisfaction Questionnaire (PSQ) at 14 days post-discharge.
Acute Care Reutilization | 30 days post-discharge
  We hypothesize that compared with usual discharge planning, PaCT patients will have lower combined rates of unplanned readmissions at 30 days post-discharge
Quality of Discharge Planning | 14 days post-discharge
  Hospital Consumer Assessment of Healthcare Providers and Systems Survey item pertaining to quality of verbal discharge communication

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Kangovi S, Mitra N, Grande D, White ML, McCollum S, Sellman J, Shannon RP, Long JA. Patient-centered community health worker intervention to improve posthospital outcomes: a randomized clinical trial. JAMA Intern Med. 2014 Apr;174(4):535-43. doi: 10.1001/jamainternmed.2013.14327. PMID 24515422